CLINICAL TRIAL: NCT00043732
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalating Study of SCIO-469 in Patients in Active Rheumatoid Arthritis Receiving Methotrexate
Brief Title: Safety Study of SCIO-469 to Treat Patients With Active Rheumatoid Arthritis Receiving Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005173
Record Dates: First submitted 2002-08-12; First posted 2002-08-14 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Scio-469
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — SCIO-469

INTERVENTIONS:
Drug: SCIO-469

SUMMARY:
The main objective of the study is to evaluate the safety and tolerability of six escalating doses of SCIO-469 in RA patients. SCIO-469 belongs to a new class of treatments that inhibit p38 kinase, a stimulatory modulator of pro-inflammatory factors including tumor necrosis factor-alpha (TNF-alpha), interleukin-1 (IL-1), and cyclooxygenase-2 (COX-2), all of which are known to contribute to both symptoms and disease progression in patients with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled, dose-escalating study will assess the safety, tolerability, efficacy, PK and pharmacodynamics of SCIO-469 in patients with active RA who also are receiving methotrexate. A total of 120 subjects will be randomly assigned and treated in one of seven dose groups with the total daily dose of SCIO-469 ranging from 0 to 180 mg. Dose groups will be staggered over four Treatment Periods. Safety and available PK data from a Treatment Period with lower dose groups will be reviewed prior to initiating higher dose groups in the next Treatment Period. Placebo subjects will be randomized in all Treatment Periods. Study drug will be taken for 30 days. Each subject will be followed for approximately 4 weeks after completing the 30-day Treatment Period. Safety will be assessed by way of physical examination, medical history, vital signs, orthostatic vital signs, chest radiograph, 12-lead electrocardiogram (ECG), clinical laboratory evaluations (including serum chemistry, hematology, qualitative urinalysis, and liver function tests), purified protein derivative test for tuberculosis, neurological tests, adverse events, and concomitant medications through out the study. Study drug will be administered for 30 days at one of the following dosage strengths; 30 mg, 60 mg, 90 mg. One group of subjects will get 60 mg for one week followed by 120 for one week followed by 180 mg for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have active rheumatoid arthritis and are receiving methotrexate
* meet the revised 1987 American Rheumatism Association (ARA) criteria for rheumatoid arthritis
* has active RA as demonstrated by 9 tender and 6 swollen joints and one of the following: C-reactive protein 1.0 mg/dL, Erythrocyte sedimentation rate (ESR) 28 mm/hour, or Morning stiffness = 45 minutes. .

Exclusion Criteria:

* Patient used etanercept, infliximab, anakinra, or an experimental biologic agent within past 3 months
* Had elevation of liver enzymes within past 6 months
* Has a history of Tuberculosis
* Vertigo, inner ear, or vestibular abnormalities
* Cancer
* HIV-positive
* Abnormal electrocardiogram
* patient has chronic or acute infection
* Multiple sclerosis, neuropathy or encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of multiple oral doses of SCIO-469 in patients with active rheumatoid arthritis (RA) who were also receiving stable doses of methotrexate (MTX).

SECONDARY OUTCOMES:
To assess the efficacy of multiple oral doses of SCIO-469 using the American College of Rheumatology (ACR) response criteria. To determine the PK of multiple oral doses of SCIO-469 in patients with active RA who are also receiving MTX.

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.